CLINICAL TRIAL: NCT00003283
Title: Phase II Study of Octreotide Treatment of Advanced, Recurrent Thymoma
Brief Title: Octreotide With or Without Prednisone in Treating Patients With Metastatic or Recurrent Thymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000066197; E-1C97
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Thymoma and Thymic Carcinoma
Keywords: invasive thymoma and thymic carcinoma; recurrent thymoma and thymic carcinoma
MeSH Terms: conditions — Thymoma | interventions — Octreotide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: octreotide acetate
Drug: prednisone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to compare the effectiveness of octreotide alone or with prednisone in treating patients with metastatic or recurrent thymoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in patients with metastatic or recurrent thymoma treated with octreotide. II. Determine the duration of remission in these patients. III. Determine the toxicity of the octreotide regimen in this population. IV. Determine the response rate, duration of remission, survival and toxicity of prednisone added to octreotide in patients with stable disease following octreotide alone.

OUTLINE: All patients receive octreotide subcutaneously three times daily for 1 month. After two courses of treatment, patients are assessed for response. Patients experiencing partial or complete response continue octreotide for a maximum of 1 year (12 courses) in the absence of unacceptable toxicity or disease progression. Patients with stable disease after 2 courses of octreotide receive daily oral prednisone in addition to octreotide for an additional 2 courses. These patients are then reevaluated and continue on octreotide plus prednisone for a maximum of 1 year in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 1 year, every 4 months for the second year, every 6 months for the next 3 years, and then annually thereafter.

PROJECTED ACCRUAL: There will be 38 patients accrued into this study over approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed invasive, recurrent, or metastatic thymoma or thymic carcinoma not amenable to potentially curative therapy Must have extensive disease defined as: - distant disease - pleural disease with or without mediastinal involvement - recurrent progressive disease in site of previous radiotherapy Measurable disease with at least one bidimensionally measurable lesion Must have octreotide scan prestudy that demonstrates activity in the area of measurable disease within 6 months prior to registration

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 3.0 mg/dL Other: No diabetes mellitus or any other complications to high dose corticosteroid therapy No acute concurrent complications such as infections Other prior malignancy(ies) must have been curatively treated and demonstrate no evidence of recurrence Not pregnant or nursing Negative pregnancy test Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior chemotherapy allowed if disease progression is demonstrated prior to study entry Endocrine therapy: Prior or concurrent corticosteroids for myasthenia gravis allowed Radiotherapy: Prior radiotherapy allowed Surgery: No postsurgical complications

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 1998-10-13 (Actual); Primary Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Ettinger, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (25):
- United States (24):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Aisner SC, Dahlberg S, Hameed MR, Ettinger DS, Schiller JH, Johnson DH, Aisner J, Loehrer PJ. Epidermal growth factor receptor, C-kit, and Her2/neu immunostaining in advanced or recurrent thymic epithelial neoplasms staged according to the 2004 World Health Organization in patients treated with octreotide and prednisone: an Eastern Cooperative Oncology Group study. J Thorac Oncol. 2010 Jun;5(6):885-92. doi: 10.1097/JTO.0b013e3181d86a30. PMID 20421818
- [Result] Loehrer PJ Sr, Wang W, Johnson DH, Aisner SC, Ettinger DS; Eastern Cooperative Oncology Group Phase II Trial. Octreotide alone or with prednisone in patients with advanced thymoma and thymic carcinoma: an Eastern Cooperative Oncology Group Phase II Trial. J Clin Oncol. 2004 Jan 15;22(2):293-9. doi: 10.1200/JCO.2004.02.047. PMID 14722038
- [Result] Loehrer PJ, Wang W, Ettinger DS, et al.: Phase II study of octreotide treatment in advanced or recurrent thymic malignancies: an Eastern Cooperative Oncology Group study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1178, 2002.